CLINICAL TRIAL: NCT03432780
Title: Randomized Phase II Clinical Study of Radiation Therapy, Hormone Therapy and Chemotherapy With Docetaxel Versus Radiation Therapy and Hormone Therapy in Patients With High-Risk Localized Prostate Cancer (Stage III and IV)"
Brief Title: Radiation-hormone and Docetaxel VS Radiation-hormone in Patients With High-Risk Localized Prostate Cancer
Acronym: QRT-SOGUG
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Collaborators: Pivotal S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: QRT-SOGUG; 2008-003554-14 (EudraCT Number)
Record Dates: First submitted 2018-01-15; First posted 2018-02-14 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Prostate Cancer Stage III; Prostate Cancer Stage IV
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Hormones; Radiotherapy

STUDY DESIGN:
Intervention Model Description: A prospective, multicenter, multidisciplinary, parallel-group, open-label study with randomized group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Docetaxel, hormone and radiation therapy (Experimental): Radiation therapy combined with weekly docetaxel (20 mg/m2) and hormone therapy.
  Interventions: Drug: Docetaxel; Biological: Hormone and radiation therapy; Radiation: Radiation therapy
- Hormone and radiation therapy (Active Comparator): Radiation therapy and hormone therapy
  Interventions: Biological: Hormone and radiation therapy; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Docetaxel
  Other Names: Taxotere
  Arms: Docetaxel, hormone and radiation therapy
Biological: Hormone and radiation therapy
Radiation: Radiation therapy

SUMMARY:
A prospective, multicenter, parallel-group, open-label, randomized, phase II Clinical Study of Radiation Therapy, Hormone Therapy and Docetaxel Versus Radiation Therapy and Hormone Therapy in Patients with High-Risk Localized Prostate Cancer (Stage III and IV) whose primary objective is determine the percentage of patients free of biochemical recurrence within 5 years of receiving a combination of radiation therapy with docetaxel associated with hormone therapy or the standard of care of radiation therapy and hormone therapy in patients with stage III and IV localized prostate cancer with a poor prognosis.

DETAILED DESCRIPTION:
Randomized Phase II Clinical Study of Radiation Therapy, Hormone Therapy and Chemotherapy with Docetaxel Versus Radiation Therapy and Hormone Therapy in Patients with High-Risk Localized Prostate Cancer (Stage III and IV) Primary Objective: To determine the percentage of patients free of biochemical recurrence within 5 years of receiving a combination of radiation therapy with docetaxel associated with hormone therapy or the standard of care of radiation therapy and hormone therapy in patients with stage III and IV localized prostate cancer with a poor prognosis.

Design: A prospective, multicenter, multidisciplinary, parallel-group, open-label study with randomized group assignment.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of adenocarcinoma of the prostate.
2. Age > 18 years.
3. Localized high-risk prostate cancer, defined as:

   * Stage III: T3 N0 M0, Gleason grade 8, 9, or 10, or
   * Stage IV: T4 N0 M0, any Gleason grade or Tx N1 M0, any Gleason grade
4. PSA > 20 ng/mL.
5. Karnofsky index ≥ 70%
6. Good bone marrow reserve, with white blood cell count > 3000/mm3, hemoglobin >9.5 g/dL and platelets > 150,000/mm3.
7. Absence of hepatic abnormality, with bilirubin values < 1.5 mg/dL and with SGOT/SGPT values up to 2 times the upper limit of normality for each site.
8. Absence of abnormality in renal function, with creatinine levels up to 2 times the upper limit of normality for each site.
9. Having given informed consent in writing.

Exclusion Criteria:

1. Previous hormone treatment during more than 3 months.
2. Previous surgical treatment, pelvic radiation therapy, or chemotherapy for the current illness.
3. Concomitant second neoplasm or history of neoplastic disease in the last 5 years, except for cutaneous basal cell carcinoma.
4. Metabolic disease or uncontrolled systemic disease.
5. Previous history of grade III-IV neuropathy (NCI CTCAE v3).
6. Psychological, social, family, or geographical conditions that may compromise compliance with or follow-up of the study.
7. Having received treatment with an investigational medicinal product during the 30 days prior to inclusion in the study.
8. Inflammatory bowel disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — prostate cancer is present only in male
Enrollment: 134 (Actual)
Dates: Start 2008-12-18 (Actual); Primary Completion 2023-11-14 (Estimated); Study Completion 2023-11-14 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients free of biochemical recurrence within 5 years of receiving a combination of radiation therapy with docetaxel associated with hormone therapy or the standard of care of radiation therapy and hormone therapy | 5 years of randomization
  Percentage of patients free of elevation of PSA by 2 ng/mL above the minimum level reached since treatment (biochemical reccurrence), calculating the at-call event, i.e., the date of last confirmatory test (Phoenix criteria).

SECONDARY OUTCOMES:
Percentage of patients with biochemical recurrence-free survival | 5 years
  The duration of survival, in months, between randomization of the patient in the study and the date of recurrence by PSA. In the remaining patients, the last available follow-up will be taken as the last control
Percentage of patients with progression-free survival | 5 years
  The duration of survival, in months, between randomization of the patient in the study and the date of recurrence by PSA, clinical manifestations or death due to disease. In the remaining patients, the last available follow-up will be taken as the last control
Percentage of patients with overall survival. | 5 years
  Defined as the time that elapses, in months, between randomization of the patient in the study and the date of death, regardless of the cause. In the remaining patients, the last available follow-up will be taken as the last control.
Clinical response rate | 5 years
  The clinical response rate: percentage of patients with partial and complete response, according to RECIST criteria.
Biochemical response rate. | 5 years
  Biochemical response rate: percentage of patients with partial and complete response, according to PSA levels.
Quality of life of the patients | screening and week 9
  Change from baseline in the Quality of Life Questionnaire C30 scale (QLQ-C30) to week 9. The QLQ-c30 has five functional scales (physical, role, cognitive, emotional, and social); three symptom scales (fatigue, pain, and nausea and vomiting); and a global health and quality-of-life scale. They are assigned values between 1 and 4 (1: nothing, 2: a few, 3: enough, 4: a lot) according to the patient's responses to the item, only in items 29 and 30 are assessed with a score from 1 to 7 (1: terrible, 7: excellent). The obtained scores are summed and standardized and gets a score between 0 and 100
Safety profile of the treatment. | 5 years
  Numbers of events evaluated according to NCI criteria CTCAE v3

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Armstrong CM, Gao AC. Drug resistance in castration resistant prostate cancer: resistance mechanisms and emerging treatment strategies. Am J Clin Exp Urol. 2015 Aug 8;3(2):64-76. eCollection 2015. PMID 26309896
- [Result] Bolla M, Collette L, Blank L, Warde P, Dubois JB, Mirimanoff RO, Storme G, Bernier J, Kuten A, Sternberg C, Mattelaer J, Lopez Torecilla J, Pfeffer JR, Lino Cutajar C, Zurlo A, Pierart M. Long-term results with immediate androgen suppression and external irradiation in patients with locally advanced prostate cancer (an EORTC study): a phase III randomised trial. Lancet. 2002 Jul 13;360(9327):103-6. doi: 10.1016/s0140-6736(02)09408-4. PMID 12126818
- [Result] Lawton CA, Winter K, Byhardt R, Sause WT, Hanks GE, Russell AH, Rotman M, Porter A, McGowan DG, DelRowe JD, Pilepich MV. Androgen suppression plus radiation versus radiation alone for patients with D1 (pN+) adenocarcinoma of the prostate (results based on a national prospective randomized trial, RTOG 85-31). Radiation Therapy Oncology Group. Int J Radiat Oncol Biol Phys. 1997 Jul 15;38(5):931-9. doi: 10.1016/s0360-3016(97)00288-5. PMID 9276357
- [Result] Kumar P, Perrotti M, Weiss R, Todd M, Goodin S, Cummings K, DiPaola RS. Phase I trial of weekly docetaxel with concurrent three-dimensional conformal radiation therapy in the treatment of unfavorable localized adenocarcinoma of the prostate. J Clin Oncol. 2004 May 15;22(10):1909-15. doi: 10.1200/JCO.2004.02.001. PMID 15143084
- [Result] Tannock IF, de Wit R, Berry WR, Horti J, Pluzanska A, Chi KN, Oudard S, Theodore C, James ND, Turesson I, Rosenthal MA, Eisenberger MA; TAX 327 Investigators. Docetaxel plus prednisone or mitoxantrone plus prednisone for advanced prostate cancer. N Engl J Med. 2004 Oct 7;351(15):1502-12. doi: 10.1056/NEJMoa040720. PMID 15470213
- [Result] Petrylak DP, Tangen CM, Hussain MH, Lara PN Jr, Jones JA, Taplin ME, Burch PA, Berry D, Moinpour C, Kohli M, Benson MC, Small EJ, Raghavan D, Crawford ED. Docetaxel and estramustine compared with mitoxantrone and prednisone for advanced refractory prostate cancer. N Engl J Med. 2004 Oct 7;351(15):1513-20. doi: 10.1056/NEJMoa041318. PMID 15470214
- [Result] Hennequin C, Giocanti N, Favaudon V. Interaction of ionizing radiation with paclitaxel (Taxol) and docetaxel (Taxotere) in HeLa and SQ20B cells. Cancer Res. 1996 Apr 15;56(8):1842-50. PMID 8620502
- [Result] Mason KA, Hunter NR, Milas M, Abbruzzese JL, Milas L. Docetaxel enhances tumor radioresponse in vivo. Clin Cancer Res. 1997 Dec;3(12 Pt 1):2431-8. PMID 9815644
- [Result] Kumar P. A new paradigm for the treatment of high-risk prostate cancer: radiosensitization with docetaxel. Rev Urol. 2003;5 Suppl 3(Suppl 3):S71-7. PMID 16985954
- See also: GLOBOCAN 2002 — https://gco.iarc.fr/
- See also: Base de datos de Mortalidad de la OMS — https://gco.iarc.fr/